CLINICAL TRIAL: NCT04507698
Title: INTense Exercise foR surVivAL Among Men With Metastatic Castrate-Resistant Prostate Cancer (INTERVAL - MCRPC): A Multicentre, Randomised, Controlled, Phase III Study
Brief Title: INTERVAL - Intense Exercise Trial for Men With Metastatic Castrate-Resistant Prostate Cancer
Acronym: INTERVAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Movember Foundation (Other); Queen's University, Belfast (Other); University of Glasgow (Other); University of Bristol (Other); University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201101
Record Dates: First submitted 2020-07-22; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer
Keywords: Metastatic; Castrate; Prostate; Cancer; Resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Exercise Arm (Experimental): If participants are placed in the Supervised Exercise Group, they will attend supervised group exercise sessions, which are individually tailored to the participants physical condition, at least once a week, every week for the first year of the study. They will be asked to exercise 3 times a week.
  Interventions: Other: Intensive Exercise Intervention
- Self-Directed Exercise Arm (No Intervention): If Participants are placed in the Self-directed Exercise Group, they will receive usual medical care (standard of care) and be asked to follow their usual exercise and lifestyle routine. They will receive supportive care in the form of newsletters, covering a variety of topics including pain management, bone health, goal setting, taking control of life, and more.

INTERVENTIONS:
Other: Intensive Exercise Intervention — INTense Exercise foR surVivAL among Men with Metastatic Castrate-Resistant Prostate Cancer (INTERVAL - MCRPC), randomised to either the supervised exercise arm or the self-directed exercise arm.
  Arms: Supervised Exercise Arm

SUMMARY:
Exercise has been established to be safe and result in improved physical function and quality of life for most individuals with cancer. However, little information exists regarding whether exercise can increase overall survival and reduce disease progression, events related to cancer spreading to the bones (e.g. bone fracture, spinal cord compression, extra radiation or surgery), and pain in patients with metastatic prostate cancer that is no longer responding to hormone therapy. The primary objective of this study is to determine if high intensity aerobic and resistance training plus psychosocial support increases overall survival compared to psychosocial support alone in prostate cancer patients.

The Movember foundation is providing support for the conduct of this study

DETAILED DESCRIPTION:
Exercise as Non-Pharmacologic Adjuvant Therapy for Prostate Cancer:

Identifying and evaluating low-toxicity adjuvant interventions that can be combined with standard therapy to improve outcomes for men with prostate cancer is a high priority and has the potential to have a large impact on the clinical and public health burden of prostate cancer. The investigators summarise briefly below promising observational, pre-clinical, and pilot clinical data that support the hypothesis that exercise improves overall survival and health-related quality-of-life (QOL) among men with advanced prostate cancer:

* Vigorous aerobic exercise after diagnosis was associated with a 60% risk of fatal prostate cancer and a 49% risk of all-cause mortality among men initially diagnosed with localised disease.
* Loading of bone inhibited growth of metastatic tumours in animal models.
* Resistance exercise and programs with both resistance and aerobic exercise improved physical function and quality-of-life in men without metastases on androgen deprivation therapy (ADT) for prostate cancer.
* Treatment-related fatigue is a common side effect in men with advanced prostate cancer and exercise may decrease fatigue and increase adherence to treatment regimens.
* New standard treatments for advanced prostate cancer cause adverse metabolic effects (e.g., weight gain, insulin resistance) that may be avoided or attenuated by exercise.

Potential mechanisms of exercise influencing prostate cancer tumour biology

Potential mechanisms by which exercise may reduce the risk of prostate cancer progression, the incidence and progression of comorbidities, treatment side effects, and overall death among men with advanced prostate cancer include:

Endocrine - Exercise influences all hormonal systems in the body with key hormones relevant to prostate cancer being testosterone, growth hormone, and insulin-like growth factor-1 (IGF-I). The androgen receptor and its transactivation by ligand are one of the most important determinants of prostate cancer progression. Measurements of serum androgens provide an important biomarker for effectiveness of androgen deprivation and prostate cancer progression. Current studies are inconclusive as to the effects of exercise on serum androgen levels. In part, these studies are limited by low patient numbers and inadequate methods for measuring testosterone levels in the low ranges seen in men on androgen deprivation therapy. This is especially true with the cyp17 inhibitors, such as Abiraterone.

Immune System, Inflammation, and Cytokines - High levels of inflammatory biomarkers are associated with an increased risk of prostate cancer-specific mortality, and exercise is known to levels of circulating inflammatory biomarkers (e.g., interleukin- 6 (IL-6)) in elderly populations. In addition, exercise may enhance natural killer cell cytotoxicity and immune surveillance, improving immune defence against prostate cancer. Further, adipokines may also have pro- or anti-oncogenic roles in angiogenesis and cell proliferation. For example, adiponectin has anti-inflammatory effects and its serum concentration is inversely correlated with adiposity. Resistin is associated with insulin resistance through AMP kinase down-regulation. It up-regulates pro-inflammatory cytokines (IL-6, tumour necrosis factor alpha (TNFα)) which act via the nuclear factor kappa-light-chain-enhancer of activated B cells (NFκb) pathway to increase transcription of proteins involved in cell proliferation, inflammation and anti-apoptosis. In addition, activation of NFκb is implicated in prostate cancer, nuclear expression being associated with nodal metastasis. IL-6 and TNFα are both elevated in the serum of patients with metastatic carcinoma compared to patients without metastases. Interestingly, both are elevated in prostate carcinoma in direct proportion to disease stage, and increases occur at the time of biochemical (PSA) disease progression.

Energy Metabolism - Exercise improves insulin sensitivity and glucose metabolism. While ADT in principle is targeting the prostate cancer tumour, the systemic treatment in patient's results in a range of alterations associated with metabolic syndrome. One of the earliest changes following ADT, within 2-6 a reduction in insulin sensitivity leading to a rise in circulating insulin (hyperinsulinemia); the rise in insulin levels precedes changes in adiposity and increased lipids, sarcopenia, and bone loss. High insulin levels are predictive of more rapid progression to CRPC, and poor prognosis. Insulin has been shown to have a direct action on prostate cancer growth and progression, and this can be inhibited by blocking insulin action. Additionally, high levels of C-peptide, a marker of insulin secretion, are associated with a more than 2-fold increased risk of prostate cancer-specific mortality. Further, over the (body mass index (BMI) >25 kg/m2) men with high C-peptide levels had a more than 4-fold increased risk of prostate cancer-specific mortality compared to normal the men with low C-peptide levels.

Body composition - Cancer and its treatments cause substantial changes in body composition with sarcopenic obesity being a common outcome. This not only results in substantial impediment to functional ability and increased cardio-metabolic risk, but also alteration of adipokine and myokine balance, which may contribute to tumour progression. Exercise increases lean muscle mass and may cause loss of fat mass, thereby improving overall body composition.

Epigenetics - Exercise can produce epigenetic modulations that may inhibit tumour cell proliferation, such as altering histone deacetylase pathways.

Telomere - Short and/or variable telomere length in the prostate is a prognostic marker among men with prostate cancer. One study among 10 men with localised prostate cancer on active surveillance reported that a lifestyle program that included moderate exercise (as the as diet, stress management, and social support) increased telomere length in blood.

Cholesterol - Epidemiological studies have suggested that high levels of cholesterol in the blood are associated with increased risk of prostate cancer and progression of prostate cancer. Exercise combined with dietary modification has been demonstrated to substantially reduce total cholesterol as the as improve the ratio of high density lipoprotein to low density lipoprotein cholesterol.

Oxidative stress - Exercise has been demonstrated to modulate oxidative stress and improve antioxidant capacity. In a pilot study at the University of California, San Francisco, men with low risk, localised prostate cancer who reported ≥3 hours/the of vigorous physical activity had modulated expression of the nuclear factor erythroid 2-related factor 2 (Nrf-2) mediated oxidative stress response pathway in their normal prostate tissue compared to men who did less exercise. Oxidative stress is hypothesized to play a significant role in the initiation and progression of prostate cancer.

As the burden of disease among men with prostate cancer advances, a rapid, significant deterioration in QOL is observed. Bone pain which is reported in up to 80% of patients with metastatic disease throughout their treatment, makes the largest single contributor to QOL deterioration in this population. Other symptoms which compromise QOL include urinary frequency, sexual dysfunction, nausea and vomiting, loss of appetite and dyspnoea. The benefits of exercise training on QOL for men with non-metastatic prostate cancer are the described, and include improvements in general QOL and also cancer-specific concerns including fatigue and sexual health. Whether exercise can improve QOL among men at the end stage of this disease is not known.

Metastatic spread of prostate cancer occurs primarily to sites in the axial skeleton including the femur, pelvis and vertebrae. Metastatic lesions, which are typically osteoblastic, lead to significant bone pain and compromised skeletal quality. Skeletal complications, such as bone fractures, orthopaedic intervention or spinal cord compression, which develop due to bone metastases, result in significant patient morbidity and compromised QOL. Furthermore, compared to those who do not experience a symptomatic skeletal related event (SSE), the occurrence of a SSE is associated with increased patient mortality. A modular multi-modal approach to exercise training involving individualised prescription of exercise to reduce the forces going through the bone has been shown to be safe and feasible in men with bony metastases and not associated with increased risk of pathological fracture. This proposal will test whether exercise training delays time to SSE as the time to progression of pain and affects measures of pain severity and opiate use. Control or relief of pain and delay or prevention of SSE are both indications for approved therapeutic agents for men with metastatic prostate cancer.

In addition to SSE and pain due to the infiltration of metastatic prostate cancer in bone, men with this disease also experience debilitating cancer-related fatigue and adverse cardio-metabolic health as a side effect of therapy. Cancer-related fatigue is a distinct phenomenon from fatigue experienced by healthy individuals and significantly health-related QOL. There are extensive data to support that exercise improves fatigue in men with a disease burden. This proposal will be the first to examine whether exercise improves or delays onset of cancer-related fatigue in men with metastatic prostate cancer.

Rationale for Focus on Metastatic Castrate-Resistant Prostate Cancer (MCRPC), our overarching objective is to determine the effect of exercise on overall survival among men with advanced prostate cancer. The investigators have chosen to restrict our study population to men with progressive MCRPC because: 1) Men with progressive MCRPC are at high risk for death within a time frame that can be feasibly tested in the setting of a RCT (median OS on treatment = 3242 to 3543 months). 2) With the proper use of stratification variables (treatment and study site), it is possible to define a homogenous study population in terms of risk of death; 3) This is the largest group of patients that can be uniformly considered to have advanced prostate cancer and thus provides the largest patient pool for recruitment while also meeting criteria 1 & 2; 4) while new therapies for MCRPC extend life, they also cause significant harm to metabolic and cardiac function and health-related QOL which may be attenuated or avoided through exercise; and 5) the investigators hypothesize that exercise will have the largest measurable effect on OS among men with documented evidence of progressing MCRPC (in contrast to men with stable M1 CRPC, non-castrate resistant disease, or non-metastatic disease).

The primary endpoint for this randomised controlled trial will be overall survival (OS). OS was chosen as the primary endpoint because it has clear biological, clinical and public health significance and is a validated endpoint for approval of new treatments among men with MCRPC. Additionally, OS data can be obtained with minimal loss to follow-up through review of medical and death records. The median OS among men with MCRPC is 3242 to 3543 months. Thus, OS is a feasible outcome to examine within the budget and timeline of the proposed study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be mCRPC. This is defined as adenocarcinoma of the prostate with systemic metastatic disease despite castrate levels of testosterone (<50 ng/dL) due to orchiectomy or LHRH agonist.

Patients must have one or more of the following to be considered mCRPC

* Metastatic Disease Progression: >20% increase in the sum of diameters of measurable lesions from the time of maximal regression or appearance of one or more new lesions.
* Bone Scan Progression: Appearance of one or more new lesions on bone scan attributable to prostate cancer.
* PSA Progression: PSA ≥2 ng/ml that has risen serially on at least two occasions, each at least one week apart (PSA1 < PSA2 < PSA3).
* Castrate levels of testosterone must be maintained while on study. Be on androgen deprivation therapy (ADT) with a GnRH agonist/antagonist or prior bilateral orchiectomy. All patients will be required to be on ADT during the study period or have had a prior bilateral orchiectomy. Men with small cell neuroendocrine tumours or features of small cell disease are not eligible.
* At enrolment, patients must fit into one of the following 5 categories:

  1. Treatment naïve for mCRPC (have not yet started approved therapies for CRPC i.e.: Abiraterone/Enzalutamide/Apalutamide/Docetaxel; less than 4 weeks on approved therapies is still considered to be treatment naïve) Or
  2. Receiving Abi/Enza/Apa for mCRPC AND responding or stable (PSA values must be stable or declining after at least 4 weeks since starting Abi/Enza/Apa for mCRPC) Or
  3. Patients with PSA progression while on Abi/Enza/Apa are eligible as long as they are asymptomatic AND there is no intent on starting chemotherapy within 6 months Or
  4. Patients treated with Docetaxel as first line therapy for mCRPC who are asymptomatic without ANY evidence of progression Or
  5. Patients may have progressed following Docetaxel first line and are now receiving treatment with Abi/Enza/Apa. These patients must absolutely be responding or stable (PSA values must be stable or declining after starting Abi/Enza/Apa treatment) and have an expected life expectancy of more than 1 year.

     * 4 weeks since last major surgery and fully recovered.
* No known contraindications to high intensity exercise, including, but not limited to: brain metastases; current congestive heart failure(New York Heart Association Class II, III or IV); serious or non-healing wound, ulcer, or bone fracture; spinal cord compromise or instrumentation due to metastatic disease; peripheral neuropathy INTERVAL Protocol Version 4.0, 19 April 2018 4

  ≥grade 3. No serious cardiovascular events within 12 months including, but not limited to, transient ischemic attack (TIA), cerebrovascular accident (CVA), or myocardial infarction (MI). Patients with a history of hypertension must be well-controlled (< 160/90) on anti-hypertensive therapy.
* Halabi Nomogram score <1951 (Risk Category rated as low or intermediate risk)
* Age ≥18 years
* Required Baseline Laboratory Values: ANC ≥ 1500/uL; Platelet count ≥ 100,000/uL; Creatinine ≤ 1.5 x upper limits of normal; Bilirubin ≤ 1.5 x upper limits of normal; AST ≤ 1.5 x upper limits of normal; Serum testosterone ≤ 50 ng/dL
* ECOG performance status 0-1
* Medical clearance by treating physician to undergo a symptom-limited cardiopulmonary exercise test and vigorous aerobic and resistance exercise training, and able to complete an acceptable cardiopulmonary exercise test.
* Exercise Coordination Centre (ECC) review and approval of subject's screening bone scan / areas with bone metastases.
* Men participating in vigorous aerobic exercise for >60 min/week or structured resistance exercise ≥2 days/week, are not eligible.
* Subject is willing and able to use technological aspects of the trial.
* The subject is fluent in the language

Exclusion Criteria:

* Previous radiographic or clinical progression (PSA progression is permitted) while on treatment with abiraterone, enzalutamide, apalutamide, or a combination.
* Previously identified small cell neuroendocrine tumours or pure small cell carcinoma of the prostate, based on a prior biopsy of the prostate.
* Brain metastases (brain imaging is not required)
* Previous and/or concurrent treatment with other anti-cancer treatments is permitted. Patients are allowed to be treated with chemotherapy during the duration of the trial. Patients who have received chemotherapy as part of initial androgen deprivation therapy for metastatic castration sensitive disease are eligible.
* Currently receiving experimental treatment with non-approved drugs at the time of enrolment. Patients must undergo a 28-day washout between last dose and screening CPET.
* Poorly controlled hypertension. During screening ≥2/3 of readings must be < 160/90, regardless of whether on a regimen of anti-hypertensive therapy or not.

If patient is currently taking hypertensive medication(s)/therapy, please indicate medication and include in the Treatment and Concomitant Medications Log (SOM: Appendix 11).

* Current congestive heart failure (New York Heart Association Class II, III or IV)
* Recent serious cardiovascular events (within 12 months) including, but not limited to, transient ischemic attack (TIA), cerebrovascular accident (CVA), or myocardial infarction (MI).
* Medical condition such as uncontrolled infection or cardiac disease that, in the opinion of the physician, would make this protocol unreasonably hazardous for the patient.
* Patients with a currently active second malignancy other than non-melanoma skin cancer. Patients are not considered to have a currently active malignancy if they have completed necessary therapy and are considered by their physician to be at <30% risk of relapse at time of assessment.
* Psychiatric illness, which would prevent the patient from giving informed consent or adhering to the study protocol.
* Serious or non-healing wound, ulcer, or bone fracture.
* Known spinal cord compromise or instrumentation due to metastatic disease in the mCRPC state. Radiation therapy for metastatic disease is allowed.
* Peripheral neuropathy ≥grade 3.
* Men participating in vigorous aerobic exercise for more than 60 minutes per week or structured INTERVAL Protocol Version 4.0, 19 April 2018 15 Resistance exercise two or more days per week (seek ECC approval before exclusion).

Experiences shortness of breath, chest discomfort, or palpitations when performing activities of daily living (patient with these symptoms can participate in the study with cardiologist clearance)

* Ongoing restriction of physical activity with physician documentation
* Has chest pain brought on by physical activity (patient can participate in the study with cardiologist clearance)
* Has developed chest pain in the past month (patient can participate in the study with cardiologist clearance)
* Moderate-to-severe bone pain (i.e., National Cancer Institute's Common Terminology Criteria for Adverse Events grade 2-3 bone pain).
* Men who do not complete the baseline lifestyle and quality-of-life questionnaires and 3-days of diet diaries or country-specific FFQ will not be eligible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male prostate cancer patients
Enrollment: 80 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 24 months
  Patients will be followed for death a minimum of 36 months after randomisation. Overall survival will be measured from the time of randomisation until death. Medical records and death certificates will be reviewed every 6 months to obtain survival status. Country-specific mortality status databases will also be searched annually; cause of death will be determined through review of medical and death records. Patients will be contacted once a year, and follow up with next of kin then alternate contact, if needed, if we do not hear from them.

SECONDARY OUTCOMES:
Disease progression | 24 months
  Progression will be determined by the treating physician, and may include any of the following, based on PCWG-3 and RECIST 1.1 criteria:
  * Bone scan: Appearance of ≥ 2 new lesions on bone scan, if bone scan >12 weeks after randomisation
  * CT/MRI: ≥ 20% increase in the sum of diameters, taking the reference as the smallest sum on study. In addition to the relative increase by 20%, the sum must also demonstrate an absolute increase >5 mm / appearance of one or more new lesions / Unequivocal progression of baseline unmeasurable lesions.
  * initiating a new therapy for MCRPC
  * Symptomatic-skeletal related event (SSE). Progression free survival will be measured from randomisation until the first of the following: first CT or bone scan documenting disease progression, initiation of a new therapy for MCRPC (clinical progression), or first SSE.
  CT Scan Progression of Non-measurable Lesions Progression will be defined based on PCWG;-3 and RECIST 1.1 as all other lesions, including
Symptomatic Skeletal Related Events | 24 months
  Time to first occurrence of SSE will be defined as the time from randomisation to documentation of any of the following (whichever occurs first) + 1 day:
  * Use of external beam radiation therapy to relieve bone pain
  * Occurrence of new symptomatic pathological bone fractures that may be vertebral or non-vertebral. Asymptomatic compression fractures detected by radiology review only will not be considered a SSE.
  * Spinal cord compression
  * Change in antineoplastic therapy to treat bone pain
  * Surgical intervention to treat bone pain
  Adverse event, concomitant medication, concomitant treatment, or survival follow-up CRFs and the participant's medical record will be the source of these findings and presented as categorical data.
Analgesic/Opiate Use | 24 months
  Analgesic/opiate use will be assessed via Brief Pain Inventory - Short Form (BPI-SF) questionnaire and the World Health Organisation (WHO) analgesic scale, and medical record review at entry with a lead-in period (<28 days). The WHO analgesic scale will be completed every three cycles (based on medical review) and BPI-SF questionnaires will be administered every three cycles until month 24, and yearly thereafter.
  BPI-SF scoring:Score: 1 - 4 = Mild Pain, Score: 5 - 6 = Moderate Pain, Score: 7 - 10 = Severe Pain.
  WHO scoring: 1 = non-opiods (e. g. acetaminophen), 2 = as necessary, mild opiods (e. g. codeine), 3 = then strong opiods (e. g. morphine or hydromorphone) until the patient is free of pain.
Metabolic Biomarkers | 24 months
  Inflammatory and cytokine systemic milieu: Serum/plasma aliquots (baseline and cycle 6) from all patient samples are intended for interrogation of a panel of markers associated with inflammation including IL1β, IL-2, IL-6, TNFα and adiponectin. Results from these investigations will be correlated with c-reactive protein and measured outcomes of exercise response and disease progression. Insulin/Glucose Metabolism: Serum aliquots (baseline and cycle 6) from all patient samples are intended for assessment of insulin levels by e.g. enzyme-linked immunosorbent assay (ELISA). Insulin sensitivity will be calculated using these fasting serum insulin values and plasma glucose determinations obtained in the additional clinical blood assessments, where the HOMA-IR method will be applied. C-peptide will also be assessed. Androgen biosynthesis: Serum aliquots from all patient samples at baseline are intended for assessment of androgen levels (Testosterone, DHT, androstenedione, DHEA, 17-hydroxy.
Physical Function | 24 months
  Physical function will be assessed using strength assessments (1RM), a cardiopulmonary exercise test (CPET) and a functional performance test (400m walk). Strength assessments will be quantified in kilograms lifted, and will be dependent upon the location and size of bone metastatic lesions present as to which tests are performed (Chest Press, Leg Press, Seated Row and Leg Extension). All strength assessments should be attempted if not contraindicated. Cardiopulmonary exercise capacity will be quantified by VO2peak (L.min and mL/(kg·min)) and workload achieved (watts) during a successful CPET (RPE ≥
Quality of Life - Patient Reported Outcome Measures | 24 months
  Symptoms will be considered independently of other outcome measures. Pain will be assessed via BPI-SF and medical record review at entry with a lead-in period (<28 days) and repeated measures will occur every three cycles. Changes occurring within 12 weeks of study initiation will be ignored in the absence of compelling evidence of disease progression. Response or progression of pain will be confirmed through repeat assessments separately by at least three weeks. Quality of life measured by the FACT-G, FACIT-Fatigue, QLQ-C30, EPIC-26, and EQ5D will be assessed every 3 cycles.

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Queens University Belfast, Belfast, Northern Ireland
  - University of Glasgow, Glasgow
  - Guy's and St Thomas's NHS Trust, London
  - University of Surrey, London

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT04507698/Prot_SAP_000.pdf